CLINICAL TRIAL: NCT05171764
Title: Feasibility and Data Collection of Dual Energy Cardiac CT on a Wide Coverage System
Brief Title: Dual Energy Cardiac CT Data Collection and Evaluation
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: 219693723
Record Dates: First submitted 2021-11-25; First posted 2021-12-29 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Coronary CTA: After the subject undergoes the standard of care, clinically indicated cardiac CT scan for diagnostic purposes, the investigational scan using the GSI Cardiac Scan Mode will be conducted utilizing the same contrast administration.
  Interventions: Device: Additional Gemstone Spectral Imaging (GSI) cardiac scan

INTERVENTIONS:
Device: Additional Gemstone Spectral Imaging (GSI) cardiac scan — After the subject undergoes the clinically prescribed cardiac Computed Tomography (CT) scan for their diagnostic purposes, the investigational Gemstone Spectral Imaging (GSI) scan will be conducted following the diagnostic CT scan utilizing the same contrast administration.

SUMMARY:
This study is intended to collect clinical feasibility data using this prototype research mode for the purposes of understanding potential clinical impact, potential limitations and strengths, and to further develop the technique through development of image reconstruction and processing approaches or identification of other areas of development required.

DETAILED DESCRIPTION:
Up to 38 subjects may be enrolled to achieve the target number of 30 evaluable subjects. Withdrawn or discontinued subjects who are enrolled and received the investigational scan, may be replaced. Subject participation will be deemed complete once the diagnostic and investigational scans are completed. A subject is considered evaluable when images and raw data from the diagnostic single energy cardiac CT scan and raw data from the investigational dual energy cardiac CT scan have been collected successfully and demonstrate a diagnostic interpretation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 50 years old undergoing routine cardiac CT imaging exam;
2. Patients that within last 12 months did not undergo medical procedures involving ionizing radiation;
3. Signed informed consent.

Exclusion Criteria:

1. Contradictions to contrast;
2. Contraindications for beta blocker;
3. BMI >30;
4. High heart rate ≥75 BPM;
5. Atrial Fibrillation;
6. Arrythmia or irregular heartbeats;
7. Pregnant women;
8. Patients lacking capacity in providing informed consent
9. Patients who did participate in prior research studies with ionizing radiation in the last 12 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled that will be undergoing a routine cardiac CT imaging scan. Subjects will be representative of the general population expected to undergo cardiac CT imaging as standard of care clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Collect Data | through study completion, an average of 1 year
  Data will be collected from the scanner for future post-processing and engineering development. There is no analysis planned at this time for the data, simply data collection.

SECONDARY OUTCOMES:
Evaluation- Likert Scale | through study completion, an average of 1 year
  Complete an image evaluation using a 5 point Likert Scale (1 - Non-Diagnostic to 5 - Excellent Image Quality), done by a qualified cardiac imaging expert.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Challman, Study Director — GE Healthcare
Locations (1):
- Zürich University Hospital, Zurich, Switzerland